CLINICAL TRIAL: NCT04854330
Title: The Acute Effect of Ketone Esters on Energy Metabolism, Cardiorespiratory Fitness and Cardiovascular Health in People With Type 2 Diabetes Mellitus.
Brief Title: Ketone Esters in T2DM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Portsmouth (Other)
Collaborators: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Principal Investigator, Ant Shepherd, Senior Lecturer in Physical Activity, Exercise and Health, University of Portsmouth
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 007
Record Dates: First submitted 2021-04-13; First posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The proposed study design will be a randomised placebo-controlled, double-blind, crossover study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Independent technician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone ester (Active Comparator): A Kme commercially available supplement will be given to the participants in the form of (R)-3-hydroxybutyl (R)-3-hydroxybutyrate (ΔG®; TΔS Ltd, UK, Oxford, UK; 0.30 ml.kg-1 body mass) and will be ingested with water and cherry-flavoured stevia in a total volume of 100 ml. Immediately following ingestion of the ketones, participants will be given 20 ml of calorie-free sparkling spring water (The Holywell Water Company Ltd, UK) in an attempt to remove any remaining flavour of the supplement.
  Interventions: Dietary Supplement: Ketone monoesters
- Placebo (Placebo Comparator): In the placebo condition, participants will consume 100 ml of water and cherry-flavoured stevia followed by the same 20 ml calorie-free sparkling spring water.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ketone monoesters — A Kme commercially available supplement will be given to the participants in the form of (R)-3-hydroxybutyl (R)-3-hydroxybutyrate (ΔG®; TΔS Ltd, UK, Oxford, UK; 0.30 ml.kg-1 body mass) and will be ingested with water and cherry-flavoured stevia in a total volume of 100 ml.
  Arms: Ketone ester
Dietary Supplement: Placebo — In the placebo condition, participants will consume 100 ml of water and cherry-flavoured stevia followed by the same 20 ml calorie-free sparkling spring water.
  Arms: Placebo

SUMMARY:
Type 2 diabetes mellitus (T2DM) reduces the ability of the body to use sugar as a fuel. As an alternative people with T2DM can use fat from the blood stream instead. Fat is a good store of energy, however, the body requires about 20% more oxygen to produce energy from fat compared to sugar. People with T2DM often have heart disease as well. This can lead to limited availability of oxygen in the heart muscle, which increases the workload of the heart and will impact on the ability to perform everyday tasks, such as walking up a flight of steps. Recently, it has been suggested that ketone esters (a sports drink that contains ketones) may be used as an alternative source of energy for people with diabetes as they are approximately 8% more efficient than fat. The investigators will assess whether these ketones can be used as a more efficient source of energy and improve how the heart works in people with T2DM. If successful, this is a relatively cheap treatment, which could be immediately implemented in people with T2DM to improve heart function and the ability to perform everyday tasks.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is a chronic and progressive metabolic disease associated with an increased prevalence of cardiovascular events, and therefore represents a significant global health concern. The aetiology of the disease is complex and involves the interaction of both non-modifiable (i.e., genetic predisposition) and modifiable (e.g., physical activity levels, diet, body mass) risk factors. Individuals with T2DM have an impaired ability to utilise glucose, the body's most efficient energy substrate (providing 2.58 ATP per molecule of oxygen), due to a decreased capacity to produce and/or utilise insulin. Consequently, there is an increased reliance on the metabolism of less efficient fuel sources, predominantly the metabolism of the free fatty acid palmitate, which produces 2.33 ATP per molecule of oxygen and thereby increases oxygen requirements by approximately 10% relative to glucose metabolism. This increased oxygen cost that manifests at rest and during exercise, increases the effort required to perform physical tasks which may discourage physical activity, further exacerbating the disease state and the prevalence of associated cardiovascular co-morbidities, and may ultimately reduce quality of life.

Whereas at high concentrations, ketone bodies are known to be toxic, at a low dose ß hydroxybutyrate, one of the most common ketone bodies produced, can be used as a metabolic substrate. Although not an efficient store of energy per se, the energy can be released at a lower O2 cost than free fatty acids, generating 2.50 units of ATP per unit of O2 consumed. Theoretically, this 7% improvement in efficiency would be of benefit to those with heart disease and diabetes. Whilst there are several studies demonstrating the theoretical benefit of this improvement in efficiency in vitro or in animal models, to date this has not been demonstrated in humans.

Sodium glucose transporter 2 (SGLT-2) inhibitors, a class of anti-hyperglycaemic agents, have been shown to suppress insulin production whilst stimulating glucagon, an action that engenders mild hyperketonaemia. Interestingly, recent trials have suggested the use of SGLT-2 inhibitors have a cardio-protective effect indicated by a significant reduction in cardiovascular related death in people with type 2 diabetes. It is hypothesised that this benefit is mediated through alternate substrate utilisation. These medications, however cannot be used for all individuals. They are not licensed for, nor are likely to be effective for people with impaired renal function, which is common among people with heart failure and diabetes. The associated risk of genital infections is over 10% even in those who have been prescribed the SGLT-2 inhibitors medication.

Exogenous ketone supplements can be ingested in the form of ketone esters and have been proven efficient in improving metabolic profile by decreasing circulating glucose and free fatty acids. More specifically a ketone monoester (Kme) supplement has been shown to provide a rapid increase in blood ß-hydroxybutyrate levels within 30 min in healthy humans. Importantly, once ingested, Kme is metabolised into ß-hydroxybutyrate, which is the isoform produced by endogenous ketogenesis. Therefore, the oral consumption of Kme may be an interesting alternative for increasing ß hydroxybutyrate and therefore improving metabolic efficiency and cardiovascular function in individuals with T2DM.

ELIGIBILITY:
Inclusion Criteria:

• HbA1c > 48 mmol/mol

Exclusion Criteria:

* they present with severe renal impairment (eGFR < 30ml/min)
* they use concomitantly GLP-1 Receptor agonists (which reduce glucagon and therefore hydroxybutyrate production);
* they currently participating in a very low calorie diet or restricted carbohydrate diet (which artificially increase endogenous ketone production);
* they present uncontrolled hypertension (systolic blood pressure > 180 mmHg);
* they have a history of myocardial infarction or cerebro-vascular events in the last 3 months;
* have a a BMI > 40 kg/m2;
* they are unable to exercise;
* they have an allergy or intolerance to ketone esters ;
* they are unable to give informed consent
* have any other serious medical condition which in the opinion of study investigators would interfere with safety or data interpretation.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-04-26 (Estimated); Primary Completion 2023-02-21 (Estimated); Study Completion 2023-02-21 (Estimated)

PRIMARY OUTCOMES:
Cardiac output | Crossover design. Assessed once on placebo and Ketone esters ~7 days apart
  Using thoracic impedance cardiography (Q-Link PhysioFlow, Manatec Ltd, Poissy, France), we will non-invasively measure stroke volume (ml/m2) and HR (b/min) to calculate cardiac output (L/min) at rest and during exercise.

SECONDARY OUTCOMES:
Fuel utilisation test | Crossover design. Assessed once on placebo and Ketone esters ~7 days apart
  Pulmonary gas exchange and ventilation will be measured non-invasively at rest (resting metabolic rate (RMR)) (Clinical Metabolic Cart, COSMED Ltd, Rome, Italy).
Exercise capacity and fuel utilisation during exercise test | Crossover design. Assessed once on placebo and Ketone esters ~7 days apart
  : In order to assess the change in fuel utilisation during exercise multiple intensities are required (i.e. rest, submaximal, i.e. below the gas exchange threshold and maximal). To assess fuel utilisation at different intensities, participants will be asked to perform a step incremental test on a cycling ergometer while breathing through a gas-exchange mask (Clinical Metabolic Cart, COSMED Ltd, Rome, Italy).
Near infrared spectrometry (NIRS) | Crossover design. Assessed once on placebo and Ketone esters ~7 days apart
  Near infrared spectrometry (NIRS) will be utilised to see if O2 extraction in the muscle changes after ketone ester ingestion and estimate changes in microvascular blood flow (Artinis Portamon, Elst, The Netherlands). This would be suggestive of an improved microvascular function and may explain changes in V ̇O2peak (i.e. exercise capacity).
Ketone concentration | Crossover design. Assessed once on placebo and Ketone esters ~7 days apart
  Human beta Hydroxybutyrate
Troponin concentration | Crossover design. Assessed once on placebo and Ketone esters ~7 days apart
  Cardiac biomarker
IL6 concentration | Crossover design. Assessed once on placebo and Ketone esters ~7 days apart
  Inflammatory biomarker
IL10 concentration | Crossover design. Assessed once on placebo and Ketone esters ~7 days apart
  Anti inflammatory biomarker
VEGF | Crossover design. Assessed once on placebo and Ketone esters ~7 days apart
  vascular endothelial growth factor

IPD SHARING:
Plan to Share IPD: Undecided